CLINICAL TRIAL: NCT03470246
Title: Personalized Intervention to Increase Physical Activity and Reduce Sedentary Behaviour in Rehabilitation After Cardiac Operations (the PACO Trial)
Brief Title: Personalized Activity Intervention in Rehabilitation After Cardiac Operations (the PACO Trial)
Acronym: PACO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: UKK Institute (Other); Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KUH5101117
Record Dates: First submitted 2018-02-28; First posted 2018-03-19 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease; Aortic Valve Stenosis; Mitral Valve Insufficiency
Keywords: Accelerometer; Aortic valve replacement; Aortic valve stenosis; Coronary artery bypass grafting; Coronary artery disease; eHealth; Interactive guidance; Mitral valve insufficiency; Mitral valve repair; Rehabilitation
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis; Mitral Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: The PACO trial is based on randomized clinical trial. Besides the standard post-operative care, the cardiac operation patients of the intervention groups will receive activity guidance during a 90-day intervention after elective coronary artery bypass grafting, aortic valve replacement or mitral valve repair. In addition, exercise guidance (short video files) and regular mobile phone contacts from physiotherapist will be provided to the intervention patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- CABG control group (No Intervention): The group of coronary artery disease patients receiving the standard postoperative rehabilitation of Kuopio and Turku university hospitals after coronary artery bypass grafting. The post-operative rehabilitation includes written and oral physical activity guidance from a physiotherapist.
- PACO intervention for CABG patients (Experimental): The group of coronary artery disease patients receiving the PACO intervention for CABG patients besides the standard postoperative rehabilitation of Kuopio and Turku university hospitals after coronary artery bypass grafting. The PACO intervention includes activity guidance (i.e. goals to improve daily steps and physical activity levels, and reduce prolonged sitting) provided to the patients with the novel combination of ExSed application, MoveSense accelerometer and cloud system. In addition, exercise guidance (short video files) and regular mobile phone contacts from physiotherapist will be included to the intervention.
  Interventions: Behavioral: PACO intervention for CABG patients
- AVR control group (No Intervention): The group of aortic valve stenosis patients receiving the standard postoperative rehabilitation of Kuopio and Turku university hospitals after aortic valve replacement. The post-operative rehabilitation includes written and oral physical activity guidance from a physiotherapist.
- PACO intervention for AVR patients (Experimental): The group of aortic valve stenosis patients receiving the PACO intervention for AVR patients besides the standard postoperative rehabilitation of Kuopio and Turku university hospitals after aortic valve replacement. The PACO intervention includes activity guidance (i.e. goals to improve daily steps and physical activity levels, and reduce prolonged sitting) provided to the patients with the novel combination of ExSed application, MoveSense accelerometer and cloud system. In addition, exercise guidance (short video files) and regular mobile phone contacts from physiotherapist will be included to the intervention.
  Interventions: Behavioral: PACO intervention for AVR patients
- MVR control group (No Intervention): The group of mitral valve insufficiency patients receiving the standard postoperative rehabilitation of Kuopio and Turku university hospitals after mitral valve repair. The post-operative rehabilitation includes written and oral physical activity guidance from a physiotherapist.
- PACO intervention for MVR patients (Experimental): The group of mitral valve insufficiency patients receiving the PACO intervention for MVR patients besides the standard postoperative rehabilitation of Kuopio and Turku university hospitals after mitral valve repair. The PACO intervention includes activity guidance (i.e. goals to improve daily steps and physical activity levels, and reduce prolonged sitting) provided to the patients with the novel combination of ExSed application, MoveSense accelerometer and cloud system. In addition, exercise guidance (short video files) and regular mobile phone contacts from physiotherapist will be included to the intervention.
  Interventions: Behavioral: PACO intervention for MVR patients

INTERVENTIONS:
Behavioral: PACO intervention for CABG patients — The PACO intervention is based on post-operative guidance to replace prolonged SB with PA in the rehabilitation of patients recovering from coronary artery bypass grafting (CABG). The guidance will be provided to the patients with the combination of ExSed smart phone application, accelerometer and cloud system. In addition, exercise guidance (short video files) and regular mobile phone contacts from physiotherapist will be provided to the intervention patients.
  Arms: PACO intervention for CABG patients
Behavioral: PACO intervention for AVR patients — The PACO intervention is based on post-operative guidance to replace prolonged SB with PA in the rehabilitation of patients recovering from aortic valve replacement (AVR). The guidance will be provided to the patients with the combination of ExSed smart phone application, accelerometer and cloud system. In addition, exercise guidance (short video files) and regular mobile phone contacts from physiotherapist will be provided to the intervention patients.
  Arms: PACO intervention for AVR patients
Behavioral: PACO intervention for MVR patients — The PACO intervention is based on post-operative guidance to replace prolonged SB with PA in the rehabilitation of patients recovering from mitral valve repair (MVR). The guidance will be provided to the patients with the combination of ExSed smart phone application, accelerometer and cloud system. In addition, exercise guidance (short video files) and regular mobile phone contacts from physiotherapist will be provided to the intervention patients.
  Arms: PACO intervention for MVR patients

SUMMARY:
The PACO trial is a randomized clinical trial conducted in Heart Centers of Kuopio and Turku university hospitals. The coronary artery disease, aortic valve stenosis and mitral valve insufficiency patients preparing for elective coronary artery bypass grafting (CABG), aortic valve replacement (AVR) or mitral valve repair (MVR) will be randomized to either intervention or control group. The specific operation groups (CABG, AVR and MVR) will be analyzed separately. The 7-day baseline measurements of sedentary behaviour (SB), physical activity (PA) and sleep will be conducted to the patients by using the RM42 accelerometer during the pre-operative month.

After the cardiac procedure is completed and the patient is moved to post-operative ward, the control group patients will begin the standard post-operative rehabilitation program of the participating hospitals (activity guidance given by a physiotherapist). Patients in the intervention groups will follow the identical program but after discharge they will also receive personalized activity guidance through the combination of ExSed smart phone application, Suunto MoveSense accelerometer and cloud system during the first 90 days of post-operative rehabilitation. Weekly evolving daily goals to replace SB with PA (daily goals for steps, moderate PA, light PA and standing, and sitting time limit) will be designed for each patient of the intervention groups. A new daily step goal will be delivered from the cloud system to the patient's smart phone in the beginning of each week of the intervention. The daily step goal of the first intervention week is based on patient's walking distance assessed by a physiotherapist in post-operative ward. The following goals will be automatically evolved in the basis of patient's personal average step count of the previous week. The MoveSense accelerometer will measure accumulated levels of SB, PA and sleep, and transmit the data to user's ExSed application with Bluetooth. With information about accumulated levels of SB and PA, the application is able to guide the patient to accomplish the predefined activity goal. The guidance and motivation will be offered with pop-up notifications and histograms (columns are fulfilled according to patient's accumulated daily activity). The researches retain a remote access to the activity data of patients in the cloud system. The ExSed application will be connected to the cloud system with internet connection.

In addition, the patients of the intervention groups will receive short video files (lasting from 1 to 3 minutes) containing exercise guidance from a physiotherapist specialized to cardiac operation patients. These videos are available on the ExSed application during the intervention. The physiotherapist will also contact each patient (by mobile phone) with structured contact form from 1 to 4 times in a month to make sure that the intervention is proceeding as designed.

ELIGIBILITY:
Inclusion Criteria:

* An eligible patient with coronary artery disease, aortic valve stenosis or mitral valve insufficiency scheduled for elective coronary artery bypass grafting, aortic valve replacement or mitral valve repair operation.
* He / she does not have any severe disease or functional limitation limiting PA (other than CVD).
* He / she is willing to wear a hip- and wrist-worn accelerometer.
* He / she is willing and capable to use a smart phone application.

Exclusion Criteria:

* He / she ends up in prolonged intensive care after cardiac operation.
* He / she has a memory disorder (i.e. Alzheimer's disease).

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2018-04-06 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in mean daily number of steps | Improvement between baseline (during the last preoperative month) and first 3 (and 12) months after discharge.
  The improvement in mean daily number of steps after 3 months from discharge. In addition, the follow-up will be continued until 12 months after discharge. The baseline values of mean daily number of steps will be determined in a 7-day accelerometer measurements conducted to the patients before the elective cardiac operation. The mean daily number of steps after the first 3 and 12 months of post-operative rehabilitation at home will be also determined in 7-day (24 h) accelerometer measurements. The raw accelerometer data will be analyzed with Mean Amplitude Deviation and Angle for Posture Estimation -algorithms to recognize the daily steps for the 7 days of which average will be calculated for each study patient.

SECONDARY OUTCOMES:
Change in mean daily accumulated total time of light PA and MVPA | Change between baseline (during the last preoperative month) and first 3 months after discharge.
  The post-operative change in patient's mean daily accumulated total time of light and moderate to vigorous physical activity.
Change in mean daily total time of sedentary behaviour (SB) | Change between baseline (during the last preoperative month) and first 3 months after discharge.
  The post-operative change in patient's mean daily total time of SB.
Change in maximal oxygen consumption | Change between the first and third months after discharge.
  The evolvement of patient's maximal oxygen consumption (VO2 peak) will be determined in 6 minute walking test, conducted to the patients twice (after 1 and 3 months) post-operatively. Only a part of the randomized patients coming from city areas of Kuopio and Turku will be included to the measurements of maximal oxygen consumption.
Improvement in self-perceived quality of life (QoL) assessed with SAQ-7 -questionnaire | Improvement between baseline (during the last preoperative month) and first 3 months after discharge.
  The improvement in patient's post-operative quality of life after 3 months of rehabilitation. The quality of life will be determined with Seattle Angina Questionnaire 7 (SAQ-7).
Improvement in self-perceived quality of life (QoL) assessed with SF-36 -questionnaire | Change between baseline (during the last preoperative month) and first 3 months after discharge.
  The improvement in patient's post-operative quality of life after 3 months of rehabilitation. The quality of life will be determined with SF-36 -questionnaire.
Improvement in self-perceived quality of life (QoL) assessed with 15 D -questionnaire | Improvement between baseline (during the last preoperative month) and first 3 months after discharge.
  The improvement in patient's post-operative quality of life after 3 months of rehabilitation. The quality of life will be determined with 15 D -questionnaire.
Improvement in self-perceived quality of life (QoL) assessed with PHQ-2 -questionnaire | Improvement between baseline (during the last preoperative month) and first 3 months after discharge.
  The improvement in patient's post-operative quality of life after 3 months of rehabilitation. The quality of life will be determined with PHQ-2 -questionnaire.
Improvement in self-perceived quality of life (QoL) assessed with Rose Dyspnea Index | Improvement between baseline (during the last preoperative month) and first 3 months after discharge.
  The improvement in patient's post-operative quality of life after 3 months of rehabilitation. The quality of life will be determined with Rose Dyspnea Index.
Incidence of major cardiovascular events | The first 12 post-operative months
  The major cardiovascular events include: all-cause mortality, any rehospitalizations due to CVD, repeat coronary revascularization, non-operational myocardial infarction and stroke. The incidence of major cardiovascular events will be monitored from the patient records of the hospitals and HILMO database during the first 12 post-operative months. In addition, patients will be asked about cardiovascular events during research telephone contact (after 12 months of rehabilitation).
Change in the accelerometer-derived portion of deep sleep | Change between baseline (during the last preoperative month) and first 3 months after discharge.
  The change in patient's deep sleep portion after cardiac operations. Deep sleep will be recognized with accelerometer attached to patient's wrist during sleep. Accelerometer will be used during 7 days.
Change in heart rate variability | Change between baseline (during the last preoperative month) and first 3 months after discharge.
  The change in the heart rate variability.

CONTACTS AND LOCATIONS:
Overall Officials: Jari Halonen, M.D.; Ph.D., Principal Investigator — Heart Center, Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasankari S, Hartikainen J, Vasankari V, Anttila V, Tokola K, Vaha-Ypya H, Husu P, Sievanen H, Vasankari T, Halonen J. Objectively measured preoperative physical activity and sedentary behaviour among Finnish patients scheduled for elective cardiac procedures: baseline results from randomized controlled trial. BMC Sports Sci Med Rehabil. 2022 Jul 16;14(1):130. doi: 10.1186/s13102-022-00522-1. PMID 35842711
- [Derived] Abraham LN, Sibilitz KL, Berg SK, Tang LH, Risom SS, Lindschou J, Taylor RS, Borregaard B, Zwisler AD. Exercise-based cardiac rehabilitation for adults after heart valve surgery. Cochrane Database Syst Rev. 2021 May 7;5(5):CD010876. doi: 10.1002/14651858.CD010876.pub3. PMID 33962483
- [Derived] Vasankari V, Halonen J, Husu P, Vaha-Ypya H, Tokola K, Suni J, Sievanen H, Anttila V, Airaksinen J, Vasankari T, Hartikainen J. Personalised eHealth intervention to increase physical activity and reduce sedentary behaviour in rehabilitation after cardiac operations: study protocol for the PACO randomised controlled trial (NCT03470246). BMJ Open Sport Exerc Med. 2019 Jul 5;5(1):e000539. doi: 10.1136/bmjsem-2019-000539. eCollection 2019. PMID 31354960